CLINICAL TRIAL: NCT04230356
Title: A Randomized Trial of Scheduled Versus Treatment Administration of Donor-Derived Viral Specific T-cells (VSTs) for Control of Viral Infections After Allogeneic Stem Cell Transplant
Brief Title: Trial of Scheduled Versus Treatment Administration of Donor-Derived Viral Specific T-cells for Viral Infections After Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Hoxworth Blood Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-1217
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Allogeneic Stell Cell Transplant; Viral Infection
MeSH Terms: conditions — Virus Diseases | interventions — Appointments and Schedules; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VSTs to Prevent (Experimental): VSTs are given through an IV infusion 21-30 days after transplant to see if the VSTs will help prevent a viral infection.
  Interventions: Biological: Viral Specific T-cells (VSTs) Scheduled
- VSTs to Treat (Experimental): VSTs will be given only if a viral infection develops.
  Interventions: Biological: Viral Specific T-cells (VSTs) Treatment

INTERVENTIONS:
Biological: Viral Specific T-cells (VSTs) Scheduled — VSTs will be infused into stem cell transplant recipients on schedule.
  Arms: VSTs to Prevent
Biological: Viral Specific T-cells (VSTs) Treatment — VSTs will be infused into stem cell transplant recipients only if viremia is detected.
  Arms: VSTs to Treat

SUMMARY:
The purpose of this research study is to learn more about the use of viral specific T-lymphocytes (VSTs) to prevent or treat viral infections that may happen after allogeneic stem cell transplant. Allogeneic means the stem cells come from another person. VSTs are cells specially designed to fight viral infections that may happen after a stem cell transplant (SCT).

Stem cell transplant reduces the body's ability to fight infections. Viral infections are a common problem after transplant and can cause significant complications. Moreover, treatment of viral infections is expensive and time consuming, with families often administering prolonged treatments with intravenous anti-viral medications, or patients requiring prolonged admissions to the hospital. The medicines can also have side effects like damage to the kidneys or reduction in the blood counts, so in this study the investigators are trying to find a better way to treat these infections.

ELIGIBILITY:
SCHEDULED ARM:

Inclusion Criteria:

* Recipient must be at least 21 days after stem cell infusion
* Clinical status must allow tapering of any steroids to < 0.5mg/kg prednisone or other steroid equivalent
* No critical illness making VST infusion hazardous

Exclusion Criteria:

* Active acute GVHD grades II-IV.
* Uncontrolled relapse of malignancy.
* Infusion of ATG or alemtuzumab within 2 weeks prior to VST infusion. Alemtuzumab levels will be collected in the second week following stem cell infusion in patients who received alemtuzumab as part of their conditioning regimen. The level must be less than or equal to 0.15 prior to infusion of VSTs. In patients with level greater than 0.15, alemtuzumab levels can be checked serially until a level ≤ 0.15 is obtained. They would become eligible for scheduled VST infusion at that point.

TREATMENT ARM

Inclusion Criteria:

* Blood adenovirus PCR ≥1,000
* Blood CMV PCR ≥ 500
* Blood EBV PCR ≥ 9,000
* Plasma BKV PCR >1,000
* Evidence of invasive adenovirus infection. Adenovirus infection will be defined as the presence of adenoviral positivity as detected by PCR or culture from one site such as stool or blood or urine or nasopharynx. Adenovirus disease will be defined as the presence of adenoviral positivity as detected by culture or PCR from more than 2 sites such as stool or blood or urine or nasopharynx.
* Evidence of invasive CMV infection, defined as pneumonitis, retinitis, colitis, hepatitis
* Evidence of EBV-associated lymphoproliferation (EBV-LPD) defined as proven EBV-LPD by biopsy or probable EBV-LPD defined as an elevated EBV DNA level in the blood associated with clinical symptoms (adenopathy or fever or masses on imaging) but without biopsy confirmation.
* Evidence of symptomatic BK virus infection, defined as hemorrhagic cystitis or BK nephropathy.
* No active acute GVHD grades II-IV
* No uncontrolled relapse of malignancy
* No infusion of ATG or alemtuzumab within 2 weeks of VST infusion.
* Clinical status must allow tapering of any steroids to < 0.5mg/kg prednisone or other steroid equivalent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Failures | 21 - 100 days after transplant
  Treatment failure is defined as EBV>100,000, BKV >100,000, CMV >5,000 or Adv >50,000 at any time post randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MBBS, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States